CLINICAL TRIAL: NCT03526510
Title: Randomized Trial of Concomitant Hypofractionated IMRT Boost Versus Conventional Fractionated IMRT Boost for Localized High Risk Prostate Cancer
Brief Title: Hypofractionated Boost vs Conventionally Fractionated Boost for Localized High Risk Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dr. Patrick Cheung (Other)
Responsible Party: Sponsor-Investigator, Dr. Patrick Cheung, Radiation Oncologist, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pHART2 RCT
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Prostate Cancer
Keywords: High Risk Prostate Cancer; Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Fractionation (Active Comparator): Using 2 sequential IMRT plans, the pelvic lymph nodes and prostate will initially be treated to 46 Gy in 23 fractions, followed by a subsequent boost to the prostate to a total dose of 78 Gy.
  Interventions: Radiation: Conventionally Fractionated versus Hypofractionated Boost
- Hypofractionation (Experimental): Using a one phase IMRT plan, the pelvic lymph nodes will be treated to a dose of 48 Gy in 25 fractions, while the prostate will be treated to a dose of 68 Gy in 25 fractions concomitantly (simulataneous integrated boost).
  Interventions: Radiation: Conventionally Fractionated versus Hypofractionated Boost

INTERVENTIONS:
Radiation: Conventionally Fractionated versus Hypofractionated Boost

SUMMARY:
Randomized trial comparing 2 external beam radiotherapy fractionation schemes in patients with localized high risk prostate cancer. Primary endpoint is acute toxicity.

DETAILED DESCRIPTION:
Patients enrolled onto this study will be randomized to one of the following treatment arms:

* Standard fractionation: Using 2 sequential IMRT plans, the pelvic lymph nodes and prostate will initially be treated to 46 Gy in 23 fractions, followed by a subsequent boost to the prostate to a total dose of 78 Gy.
* Hypofractionation: Using a one phase IMRT plan, the pelvic lymph nodes will be treated to a dose of 48 Gy in 25 fractions, while the prostate will be treated to a dose of 68 Gy in 25 fractions concomitantly (simulataneous integrated boost).

In addition, all patients receive 1.5- 3 years of androgen deprivation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained.
* Histologically confirmed diagnosis of adenocarcinoma of the prostate.
* T1-2 N0 M0, Gleason Score <= 7, PSA 20 - 100
* T1-2 N0 M0, Gleason Score 8 - 10, PSA <= 100
* T3 N0 M0, any Gleason Score, PSA <= 100

Exclusion Criteria:

* Patients with unilateral or bilateral hip replacement.
* Patients with active collagen vascular disease.
* Patients with active inflammatory bowel disease.
* Patients with previous radiotherapy to the pelvis.
* Patients with ataxia telangiectasia.
* Patients with nodal or distant metastases

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 178 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Acute Toxicity | within 3 months after starting radiotherapy
  Proportion of patients experiencing grade >=2 acute toxicity

SECONDARY OUTCOMES:
Late Toxicity | beyond 3 months of starting radiotherapy
  Proportion of patients experiencing grade >= 2 late toxicity
Biochemical Control (Phoenix Definition) | at 5 years
  Actuarial measure of patients failing biochemically (defined as PSA nadir + 2 ng/mL)
Overall Survival | at 5 years
  Actuarial measure of patients being alive

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Cheung, MD, Study Chair — Toronto Sunnybrook Regional Cancer Centre
Locations (1):
- Sunnybrook Odette Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No